CLINICAL TRIAL: NCT04878003
Title: An Open-Label, Multicenter, Phase 2 Study Assessing the Safety and Efficacy of KRT-232 or TL-895 in Janus Associated Kinase Inhibitor Treatment-Naïve Myelofibrosis
Brief Title: Study of KRT-232 or TL-895 in Janus Associated Kinase Inhibitor Treatment-Naïve Myelofibrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRT-232-114
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Primary Myelofibrosis (PMF); Post-Polycythemia Vera Myelofibrosis (Post-PV-MF); Post-Essential Thrombocythemia Myelofibrosis (Post-ET-MF)
Keywords: navtemadlin
MeSH Terms: conditions — Primary Myelofibrosis | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): KRT-232 administered orally as 240 mg once daily on Days 1-7, off treatment on Days 8-28, in 28-day treatment cycles
  Interventions: Drug: KRT-232
- Arm 2 (Experimental): TL-895 administered orally as 150 mg twice daily continuously in 28-day cycles
  Interventions: Drug: TL-895

INTERVENTIONS:
Drug: KRT-232 — KRT-232, administration by mouth
  Arms: Arm 1
Drug: TL-895 — TL-895, administration by mouth
  Arms: Arm 2

SUMMARY:
This study evaluates either KRT-232 or TL-895 in treatment naïve patients with myelofibrosis (MF)

The study will be conducted in 2 stages. Stage 1 will evaluate safety, tolerability, and efficacy of either KRT-232 (Arm 1) or TL-895 (Arm 2) in treatment naïve patients. Stage 2 will expand enrollment in Arm 1 and/or Arm 2 if expansion criteria is met.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PMF, post-PV MF or post-ET MF (WHO)
* High-risk, or intermediate-1 and 2 risk, defined by Dynamic International Prognostic System (DIPSS)
* ECOG of 0 or 1

Exclusion Criteria:

* Subjects who are positive for p53 mutation (Arm 1)
* Prior MDM2 inhibitor therapy or p53-directed therapy (Arm 1)
* Prior treatment with any JAK inhibitor
* Prior splenectomy
* Splenic irradiation within 24 weeks prior to randomization
* Prior allogeneic stem-cell transplantation or plans for allogeneic stem-cell transplant
* History of major organ transplant
* Grade 2 or higher QTc prolongation
* Major hemorrhage or intracranial hemorrhage within 24 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Spleen Volume Reduction (SVR) | 24 weeks
  The proportion of subjects achieving ≥35% SVR at Week 24 by MRI/CT (central review)

SECONDARY OUTCOMES:
Improvement in Total Symptom Score (TSS) | 24 weeks
  The proportion of subjects who have at least a 50% reduction from Baseline to Week 24 in the total symptom score as measured by the MF-SAF v4.0
Spleen Response Duration | 48 months
  Time from initial SVR of ≥35% by MRI/CT (central review) until progression
Rate of conversion from RBC transfusion dependent to independent | 24 weeks
  The proportion of subjects who convert from transfusion dependent to transfusion independent at Week 24
Overall Survival (OS) | 48 months
  Time from first dose to death from any cause
Progression free survival (PFS) | 48 months
  Time from randomization to either first occurrence of disease progression or death due to any cause

CONTACTS AND LOCATIONS:
Locations (29):
- United States (4):
  - Innovative Clinical Research Institute, Glendale, California
  - Innovative Clinical Research Institute, Whittier, California
  - Gabrail Cancer Center, Canton, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- Belarus (2):
  - Republican Scientific Practical Center of Radiation Medicine and Human Ecology, Belarus’
  - Minsk Scientific and Practice Center of Surgery, Transplantology and Hematology, Minsk
- Bulgaria (5):
  - UMHAT Georgi Stranski, Pleven
  - Medical Centre Hipokrat N, Plovdiv
  - UMHAT Sv. Ivan Rilski EAD, Sofia
  - Military Medical Academy, Sofia
  - Specialized Hospital for Active Treatment of Hematologic Diseases, Sofia
- Georgia (3):
  - JSC EVEX Hospitals, Kutaisi
  - LTD M.Zodelava Hematology Centre, Tbilisi
  - K.Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
- Mexico (4):
  - Centro de Investigacion Medica Aquascalientes (CIMA), Aguascalientes
  - Unidad de Investigacion CIMA SC, Chihuahua City
  - Centro de Investigacion Clinica de Oaxaca (CICLO), Oaxaca City
  - Sociedad de Metabolismo Y Corazon - SOMECO, Veracruz
- Poland (3):
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej Zespół Szpitali Miejskich, Katowice
  - Szpital Wojewodzki w Opolu Sp. z o.o., Oddzial Hematologii i Onkologii Hematologicznej, Opole
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku Sp. z o.o., Słupsk
- Russia (6):
  - Botkin City Clinical Hospital, Moscow
  - Republican Hospital n.a. V.A. Baranov, Petrozavodsk
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Almazov National Medical Research Center, Saint Petersburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - Samara State Medical University, Samara
- Wits Baragwanath Clinical Hematology Department, Soweto, South Africa
- City Hematology Center of Municipal Non-Profit Enterprise City Clinical Hospital #4 of Dnipro City Council, Dnipro, Ukraine